CLINICAL TRIAL: NCT06163638
Title: The Development and Evaluation of an Intergenerational Program for GRANDchildren and Their GRANDparents to Stimulate Physical Activity and Cognitive Function Using Co-creaTion
Brief Title: The Development of an Intergenerational Movement Program for Grandchildren and Their Grandparents Using Co-creation
Acronym: GRANDPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRANDPACT Project - BC-11748
Record Dates: First submitted 2022-11-08; First posted 2023-12-11 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Intergenerational Relations
Keywords: Intergenerational; Grandparents; Grandchildren; Physical activity; Cognitive functioning; Health promotion; Co-creation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: We will work with a single-case design (ABAB), where all participants will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intergenerational movement program (Experimental): This group will receive the intergenerational physical activity program. There are 4 components, which consist of an educational session for grandparents and parents (1), group-based movement sessions for grandparents and grandchildren once a week during 8 weeks (2), home-based physical activities for both grandparents and grandchildren (3) and community-based activities for both grandparents and grandchildren (4).
  Interventions: Behavioral: GRANDPACT Project

INTERVENTIONS:
Behavioral: GRANDPACT Project — To investigate whether grandparents and grandchildren are more co-physically active, have a better cognitive and physical function, psychosocial well-being, quality of the family relationship due to the intervention, we compare the intervention phase (B) with a pre phase (A), a in between period (A) and another intervention period (B)

SUMMARY:
The aim of this study is to develop, evaluate and implement an intergenerational physical activity program for grandchildren and their grandparents using co-creation focusing on the promotion of (co-)physical activity as a primary outcome and cognitive functioning, psychosocial well-being, the family relationship, expectations regarding aging and motor competence in grandparents and grandchildren as secondary outcomes.

DETAILED DESCRIPTION:
In recent years, increased attention has been devoted to intergenerational physical activity (PA) programs because they may have several benefits for children and older adults (e.g., learning skills from each other, reduction of ageism). An intergenerational PA program focusing on grandchildren and -parents in a 'standard' family setting and the combination of PA and cognitive functions is innovative and may hold potential to promote PA and improve cognitive functions in both grandchildren and their grandparents. The aim of this study is to describe the protocol of the GRANDPACT (GRANDparents and GRANDchildren improve their Physical Activity and Cognitive functions using co-creaTion) project, focusing on the development of an intergenerational PA program for grandchildren and -parents using the theoretical framework "Behaviour Change Wheel" in combination with a co-creation approach. One co-creation trajectory will be organized to develop the program, followed by an efficacy trial to refine and evaluate the program with measurements pre (at baseline), post (after 24 weeks) and follow-up (after 36 weeks) to measure the outcomes of (co-)PA, cognitive functions, psychosocial well-being, the quality of the family relationship, expectations regarding aging and motor competence in grandchildren and -parents. The outcomes will be measured using accelerometery for PA, Cambridge Neuropsychological Test Automated Battery (CANTAB) testing for cognitive functions and questionnaires for psychosocial well-being, quality of the family relationship and expectations regarding aging. Motor competence will be tested with different field tests in grandparents and grandchildren. Co-development with end-users and stakeholders during the co-creation trajectory is expected to result in an effective, attractive and feasible program. Co-PA is expected to improve PA, cognitive functions, psychosocial well-being, quality of the family relationship, motor competence and motivation to be physically active in grandchildren and -parents. Both will also have better expectations regarding aging.

ELIGIBILITY:
Inclusion Criteria for children:

* Aged between 6 and 10 years old
* Having at least 1 grandparent
* Speaking Dutch
* No serious physical, cognitive or psychiatric health problems

Inclusion Criteria for grandparents:

* Having at least 1 grandchild (aged between 6 and 10 years old)
* Speaking Dutch
* No serious physical, cognitive or psychiatric health problems

Exclusion Criteria grandparents:

- Having medical health problems (epilepsy) that can cause a risk when participating in the intervention

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change in co-PA in grandchildren and grandparents | 3 months (A: 2 weeks, B: 6 weeks, A: 2 weeks, B: 2 weeks)
  The primary outcome of the intervention is co-PA. To objectively measure co-PA, participants will be asked to wear an accelerometer (Axivity AX3) during three consecutive months. The purpose of wearing an accelerometer is to investigate whether grandchildren and their grandparents are more (co-)physically active when the intervention is adopted
Change in intensity of PA in grandchildren and grandparents | 3 months (A: 2 weeks, B: 6 weeks, A: 2 weeks, B: 2 weeks)
  In addition to the primary outcome of the intervention, which is co-PA, we would like to measure the intensity of PA during each movement session with an accelerometer (Axivity AX3)

SECONDARY OUTCOMES:
Change in general well-being in children | During 3 months, every 2 weeks
  PedsQL 8-12 General Well-Being Scale Parent report
Change in quality of the family relationship in children | 3 months, pre, between, post intervention
  Interview with parents before, during and after the intervention period
Change in general well-being in grandparents | During 3 months, every 2 weeks
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWS) - 14 items - 5-point likert scale (never, seldom, sometimes, often, always), with higher scores resulting in a higher wellbeing.
Change in quality of the family relationship in grandparents | 3 months, pre, between, post intervention
  Interview with grandparents pre, during and after the intervention
Change in cognitive functioning in grandchildren | During 3 months, every 2 weeks
  Parents will fill in the short forms of the PROMIS cognitive functioning.
  Grandchildren: 7-items on a 5-point likert scale (never, seldom, sometimes, often, always), with higher scores resulting in a better cognitive functioning
Change in cognitive functioning in grandparents | During 3 months, every 2 weeks
  Grandparents will fill in the short forms of the PROMIS cognitive functioning.
  Grandparents: 8-items on a 5-point likert scale (never, seldom, sometimes, often, always), with higher scores resulting in a better cognitive functioning
Change in physical functioning in grandparents | During 3 months, every 2 weeks
  Grandparents will fill in the short forms of the PROMIS physical functioning.
  Grandparents: 10-items on a 5-point likert scale (Without any effort, With a little effort, With some effort, With a lot of effort, Unable to do), with higher scores resulting in a better physical functioning
Change in physical functioning in grandchildren | During 3 months, every 2 weeks
  Parents will fill in the short forms of the PROMIS physical functioning.
  Grandchildren: 7-items on a 5-point likert scale (Without any effort, With a little effort, With some effort, With a lot of effort, Unable to do), with higher scores resulting in a better physical functioning
Increasing WHO themes in grandparents | During 3 months, every 2 weeks
  We ask grandparents if they did exercises focusing on condition, coordination, strength, balance and flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Cardon, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No